CLINICAL TRIAL: NCT06877078
Title: The Effect of Information About Constipation Via a Podcast for Patients Prior to Planned Orthopaedic Surgery - a Randomised Controlled Trial.
Brief Title: Effect of Pre-Surgery Constipation Podcast: A RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Appel, Research nurse, Central Jutland Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1-16-02-6-25
Record Dates: First submitted 2025-03-07; First posted 2025-03-14 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Constipation; Orthopedic Disorder
Keywords: podcast; patient information; constipation; orthopedic surgery
MeSH Terms: conditions — Constipation; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Patients cannot be blinded to whether they receive access to the podcast but will be blinded to the study hypothesis. They will be informed that the study compares two types of preoperative information on constipation. Staff involved in recruitment will be blinded to randomisation, which will be carried out using the secure online system REDCap, and researchers conducting the analyses will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Podcast Group (Experimental): Participants in the experimental group will in addition to the standard information also receive a podcast.
  The standard information is provided by a nurse at the preoperative consultation. Patients also receive a card with access to an online platform with information about constipation, the specific surgery, preparations for surgery, and the period after surgery.
  Interventions: Behavioral: Constipation information via Podcast
- Control Group (No Intervention): Participants in the control group will receive the standard information. The information is provided by a nurse at the preoperative consultation. Patients also receive a card with access to an online platform with information about constipation, the specific surgery, preparations for surgery, and the period after surgery.

INTERVENTIONS:
Behavioral: Constipation information via Podcast — The podcast is 30 minutes long, and includes information on constipation explained by a gastroenterologist specialised in defecation disorders, as well as patients' experience with constipation after surgery.
  The podcast is developed in collaboration with Silkeborg Regional Hospital and the Central Denmark Region's Centre for Competence Development.
  Patients will get access to the podcast after randomisation, and will be able to listen to it throughout the study period.
  Arms: Podcast Group

SUMMARY:
In this study, the investigators will evaluate the effect of a podcast on constipation on the number of patients with constipation. It is hypothesised that the podcast on constipation, will prevent constipation in the period leading up to and after surgery.

This is a randomised controlled trial. The population of the study will consist of patients with planned orthopaedic surgery (knee, hip, shoulder, and back) at the Elective Surgery Centre, Silkeborg Regional Hospital. The sample of the study will consist of patients 18 years or older, who are able to understand, read and write Danish, has an email address, has access to and is able to navigate a computer, tablet or smartphone, does not have severe hearing loss, does not have cognitive dysfunction or other mental illness that would make participation difficult, is not participating in other trials at the Elective Surgery Centre, is not diagnosed with a gastrointestinal condition (Crohns, Colitis ulcerosa or celiac disease), and does not previously have received a colostomy or ileostomy.

Patients will be randomised to either a control group or an intervention group. Both groups will receive the standard information at the preoperative consultation and after randomisation. The intervention group will also receive a podcast.

The study will collect data using an online questionnaire, that includes The ROME IV Diagnostic Criteria for functional constipation and "The Patient Assessment of Constipation Quality of Life (PAC-QOL)". Data will be collected at 4 times: (1) after the preoperative consultation (baseline), (2) 1-2 days prior to surgery, (3) 1 week after surgery, and (4) 4 weeks after surgery.

DETAILED DESCRIPTION:
Objective:

Primary aim: to evaluate the effect of a podcast on the number of patients with constipation at admission to surgery.

Secondary aim: to evaluate the effect of a podcast on the number of patients with constipation in the period after surgery.

Method: This is a randomised controlled trial, which will be conducted at the Silkeborg Regional Hospital, Denmark, between March and October 2025.

The study population will include patients scheduled for knee, hip, shoulder, and back surgery at the Elective Surgery Centre, Silkeborg Regional Hospital. The study population will consist of patients 18 years or older, who are able to understand, read and write Danish, has an email address, has access to and is able to navigate a computer, tablet or smartphone, does not have severe hearing loss, does not have cognitive dysfunction or other mental illness that would make participation difficult, is not participating in other trials at the Elective Surgery Centre, is not diagnosed with a gastrointestinal condition (Crohns, Colitis ulcerosa or celiac disease), and does not previously have received a colostomy or ileostomy.

Sample size: Based on calculations, 600 patients are needed to achieve 80% power at a 5% significance level, assuming 30% constipation in the control group and 10 percentage points fewer in the intervention group (ROME IV criteria).

Eligible participants will be randomised into a control group and an intervention group. Both groups will receive the standard information related to their respective surgeries. The intervention group will however also be receiving a podcast about constipation in relation to surgery. The podcast is 30 minutes long, and includes information on constipation explained by a gastroenterologist specialised in defecation disorders, as well as patients' experience with constipation after surgery. The podcast is developed in a collaboration between Elective Surgery Centre, Medical Diagnostic Centre (Silkeborg Regional Hospital) and the Central Denmark Region's Centre for Competence Development.

The outcomes are measured using online questionnaires at (1) baseline after preoperative consultation (2-6 weeks before surgery), (2) 1-3 days before surgery, (3) 1 week after surgery, and (4) 4 weeks after surgery. Primary and secondary outcome is the prevalence of constipation measured using questionnaires with ROME IV criteria. Questionnaires will also be used to collect data on quality of life (The Patient Assessment of Constipation Quality of Life (PAC-QOL)), use of laxatives (frequency and type), education level, employment, living situation, use of the standard patient information and its usefulness, and use of the podcast and its usefulness. Data will also be collected from patient records using The Region of Central Denmark's data warehouse. This will be data on hospitalisations and length of stay, rehospitalisation, type of surgery, diagnoses, contact with general practitioner, and contact with the clinic due to issues with bowel movements.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years or older.
* Has a scheduled back, shoulder, knee, or hip operation at the Elective Surgery Centre
* Is able to read, speak and understand Danish.
* Has an email address and gives consent to contact via email
* Has access to and is able to navigate a computer, tablet or smartphone

Exclusion Criteria:

* Is unable to listen to the podcast, due to severe hearing loss.
* Is affected by cognitive dysfunction or mental illness that makes participation difficult.
* Is participating in other trials at the Elective Surgery Centre.
* Is diagnosed with a gastrointestinal condition, this being Crohns, Colitis ulcerosa, or celiac disease.
* Has previously received a colostomy or ileostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-17 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
ROME IV Diagnostic Criteria for functional constipation | Measured at baseline (after preparatory consultation) and 1-3 days prior to surgery.
  The ROME IV criteria consists of 6 diagnostic criteria. To diagnose constipation using ROME IV criteria in this study, two or more of the criteria must have been fulfilled the last 3 months or since last measured.

SECONDARY OUTCOMES:
The Patient Assessment of Constipation Quality of Life (PAC-QOL) | Measured at baseline (after preparatory consultation), 1-3 days prior to surgery, and 1 week and 4 weeks after surgery.
  The Patient Assessment of Constipation Quality of Life is a questionnaire that measures quality of life of patients with constipation. It contains 28 items grouped into 4 subscales covering: Worries and concerns (11 items), Physical discomfort (4 items), Psychosocial discomfort (8 items), and Satisfaction (5 items). A 5-point Likert response scale, ranging from 0 (Not at all / None of the time) to 4 (Extremely / All of the time), is used over a 2-week recall period. Minimum score: 0 (none of the time), maximum score 112 (all of the time/extremely).
ROME IV Diagnostic Criteria for functional constipation | Measured at baseline (after preparatory consultation) and 1 week and 4 weeks after surgery.
  The ROME IV criteria consists of 6 diagnostic criteria. To diagnose constipation using ROME IV criteria in this study, two or more of the criteria must have been fulfilled the last 3 months or since last measured.
Number of hospitalizations after surgery | 30 days and 6 months after surgery
  Number of hospitalizations after surgery
Number of contacts to general practitioner after surgery | 30 days and 6 months after surgery
  Number of contacts to general practitioner after surgery
Number of outpatient visits after surgery | 30 days and 6 months after surgery
  Number of outpatient visits after surgery (all and contact to surgery department and gastroenterology department)

OTHER OUTCOMES:
Use of podcast and information material, and the usefulness of these. | Measured 1-3 days prior to surgery, and at 1 week and 4 weeks after surgery.
  In the online questionnaire, all patients will be asked about their use of the information an if they found it useful.
  The intervention group will also be asked if they have listened to the podcast, and if they found it useful.
Use of laxantia, frequency (regularly or as needed) and type. | Measured at baseline, 1-3 days prior to surgery, and at 1 week and 4 weeks after surgery.
  In the online questionnaire patients will be asked whether they use laxantia, and if so what type and how often (regularly or as needed).
Days of hospitalization after surgery | From time for admission to surgery to discharge
  Days of hospitalization after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Weiling Appel, Ph.d., Principal Investigator — Regional Hospital Central Jutland, Medical Diagnostic Centre
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No